CLINICAL TRIAL: NCT01357707
Title: Clinical-genetic Investigations in Children With Early Infantile Epilepsies
Status: Completed | Type: Observational
Sponsor: Markus Schuelke, M.D. (Other)
Collaborators: Mainz University (Other); University of Ulm (Other); Ludwig-Maximilians - University of Munich (Other); University of Kiel (Other)
Responsible Party: Sponsor-Investigator, Markus Schuelke, M.D., Prinicpal investigator, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: EA1_215_08; SFB 665 TP C4 (Other Grant/Funding Number: Deutsche Forschungsgemeinschaft)
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Epilepsy; Seizures, Infantile
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA isolated from blood cells or from saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- West Syndrome (idiopathic): Patients with idiopathic infantile seizures
  Interventions: Genetic: DNA preparation

INTERVENTIONS:
Genetic: DNA preparation — Taking blood or saliva from the patient to prepare DNA therefrom

SUMMARY:
The project strives to discover novel genetic defects that cause monogenic epilepsy or that genetically modify a preexisting epileptic phenotype. Our main aim is to find genetic causes for the idiopathic West Syndrome (infantile seizures) that are not caused by known cerebral malformation, lissencephaly or metabolic disorders and which have a comparatively benign prognosis.

The investigators hypothesize that mutations in genes coding for ion channels or genes that modify the action of ion channels might be causative.

For that the investigators will perform a sequence analysis of the coding exons of a large set of genes in all recruited patients and verify found mutations in their parents.

ELIGIBILITY:
Inclusion Criteria:

* Hypsarrhythmia in the first year of life
* Infantile seizures in the first year of life
* Freedom of seizures at the age of 5 years

Exclusion Criteria:

* brain malformation
* metabolic disorder
* intracranial hemorrhage
* lissencephaly

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with infantile seizures without brain malformations, metabolic disorders of lissencephaly who had a good outcome and are seizure free (with or without AEDs) after the age of 5 years.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2010-07; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Discovery of a pathogenic mutation in an ion channel gene | 4 weeks after taking of the DNA specimen

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Universitätsmedizin, Berlin, Germany